CLINICAL TRIAL: NCT00953368
Title: Effect of Remote Ischemic Preconditioning on Cognitive Function After Off-Pump Coronary Artery Bypass Graft
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: In-Cheol Choi, professor, Asan Medical Center, Department of Anesthesiology and Pain Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RIPC-3862
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Ischemic Heart Disease
Keywords: remote ischemic preconditioning; cognitive function; off-pump coronary artery bypass graft
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remote ischemic preconditioning (Active Comparator): Remote ischemic preconditioning will be induced by four 5-min cycles of upper limb ischemia and 5-min reperfusion with a blood-pressure cuff inflated to 200 mmHg and be performed before and after the coronary anastomosis
  Interventions: Procedure: remote ischemic preconditioning
- control (Placebo Comparator): sham placement of a blood-pressure cuff around the upper limb without inflation
  Interventions: Procedure: remote ischemic preconditioning

INTERVENTIONS:
Procedure: remote ischemic preconditioning — Remote ischemic preconditioning will be induced by four 5-min cycles of upper limb ischemia and 5-min reperfusion with a blood-pressure cuff inflated to 200 mmHg and be performed before and after the coronary anastomosis

SUMMARY:
The aim of this study is to evaluate the effects of remote ischemic preconditioning on cognitive function in patients undergoing off-pump coronary artery bypass graft.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective off-pump coronary artery bypass graft surgery

Exclusion Criteria:

* Emergency operation
* Preoperative use of inotropic drugs or mechanical assistant device
* Ejection fraction less than 30%
* Combined operation using CPB such as valve surgery
* Previous psychiatric and neurologic disorder
* Inability to perform the cognitive function test

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2009-10; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
cognitive function | preoperative, 1 week and 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: In-Cheol Choi, professor, Principal Investigator — Asan Medical Center, Department of Anesthesiology and Pain Medicine
Locations (1):
- Department of Anesthesiology and Pain Medicine, University of Ulsan, College of Medicine, Asan Medical Center, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Van Dijk D, Jansen EW, Hijman R, Nierich AP, Diephuis JC, Moons KG, Lahpor JR, Borst C, Keizer AM, Nathoe HM, Grobbee DE, De Jaegere PP, Kalkman CJ; Octopus Study Group. Cognitive outcome after off-pump and on-pump coronary artery bypass graft surgery: a randomized trial. JAMA. 2002 Mar 20;287(11):1405-12. doi: 10.1001/jama.287.11.1405. PMID 11903027